CLINICAL TRIAL: NCT01344395
Title: Local Infiltration Analgesia in Total Hip Arthroplasty - Efficacy of Multiple Bolus Injections With Ropivacaine and Ketorolac
Brief Title: Use of Local Infiltration Analgesia Following Total Hip Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Lundbeck Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009-016445-25
Record Dates: First submitted 2010-04-09; First posted 2011-04-29 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Pain, Postoperative; Pain
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Ropivacaine; Ketorolac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RK-group (Experimental)
  Interventions: Drug: ropivacaine and ketorolac
- K-group (Active Comparator)
  Interventions: Drug: Ketorolac

INTERVENTIONS:
Drug: ropivacaine and ketorolac — The RK-group receives four intra-articular injections via catheter with a total volume of 40 ml (380 mg ropivacaine and 60 mg ketorolac) combined with 4 intravenous injections of saline during 24 hours postoperatively
  Arms: RK-group
Drug: Ketorolac — The K-group receives four intra-articular injections via catheter with a total volume of 40 ml saline combined with 4 intravenous injections of ketorolac (total 60 mg) during 24 hours postoperatively
  Arms: K-group

SUMMARY:
The primary aim of this study is to evaluate if multiple postoperative administrations with a solution of ropivacaine, ketorolac and epinephrine into the operating field through a catheter would affect morphine consumption. Secondary end-points are pain intensity, side effects and length of stay.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for total hip arthroplasty
* Patients > 18 years of age
* Signed written informed consent
* Spinal anaesthesia

Exclusion Criteria:

* Allergy towards study drugs
* Rheumatoid arthritis
* Body Mass Index > 35 (severe obesity)
* Pregnancy or nursing women
* Regular opioid use
* Patients who can not read or understand danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-03; Primary Completion 2011-06 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Morphine consumption | 24 hours postoperatively
  Cummulative morphine comsumption postoperatively

SECONDARY OUTCOMES:
Pain intensity | 24 hours postoperatively
  Pain intensity measured on the visual analog scale (VAS) at rest and during walking
Postoperative nausea | 24 hours postoperatively
  Number of episodes of nausea measured on a 3 points rating scale (mild, moderate and severe)

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Søballe, Professor, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark